CLINICAL TRIAL: NCT06762639
Title: Evaluating the Effect of a Sleep Prehabilitation Intervention: A Single-blind Randomized Trial
Brief Title: Improving Patient Sleep Prior to Elective Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 24-5450
Record Dates: First submitted 2024-12-19; First posted 2025-01-07 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Surgery
Keywords: Sleep; Randomized trial; Prehabilitation; Surgical recovery

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Prehabilitation (Active Comparator): Prehabilitation at UHN's Prehabilitation Program includes assessment of patients' function followed by individualized health optimizing intervention including: exercise, nutritional support, psychosocial support, education, smoking cessation support, and/or medical care.
  Interventions: Behavioral: Standard of Care Prehabilitation
- Personalized Sleep Prehabilitation (Experimental): Sleep prehabilitation will consist of usual care prehabilitation (exercise, nutritional support, psychosocial support, education, smoking cessation support, and/or medical care) with the addition of sleep support. This support will consist of:
  * Brief behavioural treatment for insomnia
  * Sleep hygiene
  * Behaviour change support (e.g., goal-setting, use of a wearable tracker to modify behaviour)
  Interventions: Behavioral: Personalized Sleep Prehabilitation (PSP)

INTERVENTIONS:
Behavioral: Personalized Sleep Prehabilitation (PSP) — Sleep prehabilitation will consist of usual care prehabilitation (exercise, nutritional support, psychosocial support, education, smoking cessation support, and/or medical care) with the addition of sleep support. This support will consist of:
  * Brief behavioural treatment for insomnia
  * Sleep hygiene
  * Behaviour change support (e.g., goal-setting, use of a wearable tracker to modify behaviour)
  Arms: Personalized Sleep Prehabilitation
Behavioral: Standard of Care Prehabilitation — Exercise, nutritional support, psychosocial support, education, smoking cessation support, and/or medical care delivered by regulated health professionals included Kinesiologists, Dietitians, Clinical Psychologists, etc.
  Arms: Standard of Care Prehabilitation

SUMMARY:
The goal of this clinical trial is to learn if changing sleep behaviour can improve sleep health in patients undergoing prehabilitation before elective surgery. Prehabilitation is the use of exercise, nutrition, and psychological support before surgery to improve recovery from surgery.

The main questions it aims to answer are:

Does changing sleep behaviour improve sleep before surgery? Does changing sleep behaviour improve recovery after surgery?

Researchers will compare participants who receive sleep support with participants who do not receive sleep support to see if it improves sleep health and recovery from surgery.

Participants will be asked to attend 4 meetings with the research team to learn how they can improve their sleep. They will use questionnaires, a diary, and a wearable tracker to record their sleep.

DETAILED DESCRIPTION:
Sample Size: N = 154

Study Population: Patients participating in UHN's Prehabilitation Program. Participants will be excluded if they are participating in prehabilitation entirely remotely (i.e., no in-person visits), have an existing sleep disorder, are a shift worker, have travel plans outside of usual time zone, or have a cognitive disability that limits answering questionnaires or adhering to the intervention.

Study Design: Randomized trial with outcome assessors blinded to group allocation.

Primary Objective: Measure the effect of a personalized sleep prehabilitation (PSP) in addition to standard of care prehabilitation on participant sleep health compared to standard of care prehabilitation alone.

Secondary Objective: To measure the effect of the PSP versus standard of care prehabilitation on other outcomes including clinical outcomes, patient-reported outcomes, and physical fitness.

Endpoints of the study: Self-reported sleep health via the Pittsburgh Sleep Quality Index (PSQI; primary outcome). Other sleep health outcomes include the insomnia severity scale (ISI), STOP-BANG questionnaire, Restless Leg Syndrome Diagnostic Index, sleep diary, Global Sleep Assessment Questionnaire (GSAQ), and sleep self-efficacy scale. Clinical outcomes include hospital length of stay and surgical complications. Anthropometric and physical fitness outcomes include: body mass index, bioelectrical impedance analysis (lean mass and fat mass), waist circumference, muscular fitness, aerobic fitness, and functional capacity. Device measured outcomes include sleep, physical activity, resting heart rate, and heart rate variability via a wrist-worn activity tracker.

Analysis: Descriptive statistics will be used to characterize participant characteristics. The primary analysis will be an ANCOVA to detect significant differences in PSQI between groups at the preoperative timepoint while controlling for baseline scores. The secondary analysis will be a linear mixed effect model to derive point estimates for effectiveness markers (primary and secondary) at each timepoint, comparing between- and within- group differences at each timepoint. Means and 95% CI will be reported.

Impact: The proposed study will be the first to explore the effect of a PSP in addition to standard-of-care prehabilitation service on sleep health.

ELIGIBILITY:
Inclusion Criteria:

* surgery date (or expected date) is ≥ 4 weeks and ≤ 12 weeks year from the time of consent
* currently sleep < 7 hours of sleep on most nights in the past month
* consistently have a sleep latency > 30 minutes
* consistently wake up throughout the night
* consistently wake up earlier than intended
* experience daytime sleepiness

Exclusion Criteria:

* have an existing diagnosed sleep disorder that is poorly managed or requires referral to a sleep clinician
* are currently a shift worker (work schedule outside of 7am-6pm).
* have plans to travel 3 or more hours outside of their usual time zone
* do not have English proficiency
* have a cognitive disability that significantly limits ability to respond to screening questions as this will impact ability to answer questionnaires and adhere to the intervention (if applicable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | Administered baseline, one week before surgery, and 45 days after surgery
  The PSQI is a self-report measure of sleep quality among seven subscales including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction. The scale's validity and reliability has been determined among clinical and older adult populations.
  For reporting, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (min: 0 and max: 21). Higher scores indicate worse sleep quality.
  Time to completion is 5-10 minutes.

SECONDARY OUTCOMES:
Sleep self-efficacy scale | Baseline, 1 week presurgery, 45 days after surgery.
  Self reported questionnaire measuring confidence in one's ability to change sleep behaviour.
  This scale contains 13 items scored 1-5 (min: 13, max: 65). Greater scores indicate more sleep self-efficacy.
Sleep diary - Sleep duration | Baseline, presurgery, 45 days after surgery
  Self-reported by the participant in the sleep diary each day for 1 week.
Sleep diary - Sleep efficiency | Baseline, presurgery, 45 days after surgery
  Time in bed and sleep duration are self-reported by the participant in the sleep diary each day for 1 week. Sleep efficiency is calculated as sleep duration/time in bed and expressed as a percentage.
Sleep diary - Sleep latency | Baseline, presurgery, 45 days after surgery
  Self-reported by the participant in the sleep diary each day for 1 week.
Sleep diary - Sleep quality | Baseline, presurgery, 45 days after surgery
  Self-reported by the participant in the sleep diary each day for 1 week using a 5-pt Likert scale ranging from "Very poor" to "Very good" (scored 0-4). Higher scores indicate better quality sleep.
Wrist-worn actigraphy - Sleep duration | Baseline, presurgery, 45 days after surgery
  All participants will be provided with a Fitbit Inspire 3, a small non-intrusive and waterproof device that uses actigraphy to measure orientation and movement and uses photoplethysmography (PPG) to detect periodic changes in blood flow beneath the sensor; thereby measuring changes in heart rate. This device is worn like a wrist-watch. The activity tracker measures sleep-wake activity to measure sleep duration expressed in minutes.
Wrist-worn actigraphy - Sleep latency | Baseline, presurgery, 45 days after surgery
  All participants will be provided with a Fitbit Inspire 3, a small non-intrusive and waterproof device that uses actigraphy to measure orientation and movement and uses photoplethysmography (PPG) to detect periodic changes in blood flow beneath the sensor; thereby measuring changes in heart rate. This device is worn like a wrist-watch. The activity tracker measures sleep-wake activity to measure sleep latency expressed in minutes.
Wrist-worn actigraphy - Sleep efficiency | Baseline, presurgery, 45 days after surgery
  All participants will be provided with a Fitbit Inspire 3, a small non-intrusive and waterproof device that uses actigraphy to measure orientation and movement and uses photoplethysmography (PPG) to detect periodic changes in blood flow beneath the sensor; thereby measuring changes in heart rate. This device is worn like a wrist-watch. The activity tracker measures sleep-wake activity to measure time in bed and time spent sleeping to compute sleep efficiency expressed as a percentage.
Wrist-worn actigraphy - Resting heart rate | Baseline, presurgery, 45 days after surgery
  All participants will be provided with a Fitbit Inspire 3, a small non-intrusive and waterproof device that uses actigraphy to measure orientation and movement and uses photoplethysmography (PPG) to detect periodic changes in blood flow beneath the sensor; thereby measuring changes in heart rate. This device is worn like a wrist-watch. The heart rate monitor will measure resting heart rate (bpm) a metric of overall fitness and autonomic nervous system function. Participants will be provided with setup instructions at their baseline appointment and receive ongoing support for the use of their tracker.
Wrist-worn actigraphy - Heart rate variability | Baseline, presurgery, 45 days after surgery
  All participants will be provided with a Fitbit Inspire 3, a small non-intrusive and waterproof device that uses actigraphy to measure orientation and movement and uses photoplethysmography (PPG) to detect periodic changes in blood flow beneath the sensor; thereby measuring changes in heart rate. This device is worn like a wrist-watch. The heart rate monitor will measure heart rate variability, a metric of overall fitness and autonomic nervous system function. Participants will be provided with setup instructions at their baseline appointment and receive ongoing support for the use of their tracker.
Wrist-worn actigraphy - Light intensity physical activity | Baseline, presurgery, 45 days after surgery
  All participants will be provided with a Fitbit Inspire 3, a small non-intrusive and waterproof device that uses actigraphy to measure orientation and movement and uses photoplethysmography (PPG) to detect periodic changes in blood flow beneath the sensor; thereby measuring changes in heart rate. This device is worn like a wrist-watch. The actigraphy will measure light intensity physical activity reported in minutes.
Wrist-worn actigraphy - Moderate-vigorous physical activity | Baseline, presurgery, 45 days after surgery
  All participants will be provided with a Fitbit Inspire 3, a small non-intrusive and waterproof device that uses actigraphy to measure orientation and movement and uses photoplethysmography (PPG) to detect periodic changes in blood flow beneath the sensor; thereby measuring changes in heart rate. This device is worn like a wrist-watch. The actigraphy will measure moderate-vigorous intensity physical activity reported in minutes.
Physical Fitness - Body mass index | Baseline, presurgery, 45 days after surgery
  A kinesiologist will measure height and weight to calculate body mass index expressed in in kg/m^2
Physical Fitness - Body fat % | Baseline, presurgery, 45 days after surgery
  A kinesiologist will measure body fat percentage with a mBCA 514 (Seca, Hamburg, Germany)
Physical Fitness - Grip strength | Baseline, presurgery, 45 days after surgery
  A kinesiologist will measure grip strength using a handgrip dynamometer
Physical Fitness - Six minute walk test | Baseline, presurgery, 45 days after surgery
  A kinesiologist will measure aerobic fitness using a six-minute walk test on a 60m track.
Surgical complications | Up to 45 days after surgery
  Surgical complications will be extracted from participant medical records.
Hospital length of stay | Up to 45 days after surgery
  Hospital length of stay will be extracted from participant medical records.
Discharge destination | Up to 45 days after surgery
  Discharge destination will be extracted from participant medical records.
Readmission to the hospital | Up to 45 days after surgery
  Readmissions will be extracted from participant medical records
PROMIS 29+2 | Baseline, presurgery, 45 days after surgery
  The Patient-Reported Outcomes Measurement Information System (PROMIS) is a set of person-centred measures that evaluates physical, mental, and social health. The PROMIS 29+2 Profile v2.1 (PROPr) will be administered. The PROMIS instruments have been used and validated extensively in clinical
  There are 31 questions answered using a Likert scale from 1-5. Each domain (physical function, anxiety, depression, cognitive function, sleep disturbance, fatigue, social activity, and pain) has 2-4 items. Higher score is more of that concept. Raw scores are converted into T scores. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10.
  Time to completion: 5-10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Santa Mina, PhD, Principal Investigator — University Health Network, Toronto; Ian Randall, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol may be shared with publication. All other data available on reasonable request.
Access Criteria: Stakeholders may access the data upon reasonable request. Mechanism and agreement of access will be determined at the time of the request.

REFERENCES:
- [Derived] Sibley D, Randall I, Culos-Reed SN, Slepian PM, Singh M, Mina DS. Evaluating the Effect of a Sleep Prehabilitation Intervention in Patients Awaiting Elective Surgery: Protocol for a Single-Blind Randomised Trial. J Sleep Res. 2025 Aug 30:e70173. doi: 10.1111/jsr.70173. Online ahead of print. PMID 40884156
- See also: Prehabilitation Program — https://www.uhn.ca/Surgery/Clinics/Prehabilitation_Program